CLINICAL TRIAL: NCT03787862
Title: Investigation of the Use of Hyperspectral Imaging in Foot Surgery Patients
Acronym: HSI
Status: Withdrawn | Type: Observational
Why Stopped: PI No longer with the University
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HSI in Foot Surgery
Record Dates: First submitted 2014-06-13; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Foot Ulcers; Osteomyelitis; Amputation
Keywords: Foot ulcers; Foot Surgery; Hyperspectral imaging
MeSH Terms: conditions — Foot Ulcer; Osteomyelitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hyperspectral Imaging (HSI): Patients scheduled for foot surgery will be imaged using the HSI device. Data will be gathered from the electronic medical record for one year to determines the outcomes of the surgery, any complications, re-hosptializations, re-ulcerations or amputation.

SUMMARY:
To investigate novel advanced imaging techniques (hyperspectral imaging) that could enable clinicians to determine the degree and effectiveness of blood flow to tissues during surgery.

There are a number of disorders where blood flow is inadequate to provide nutrients and oxygen to tissues. Under some circumstances, surgery is required to either improve the blood flow or remove tissues that are poorly perfused. In other cases, occlusion of the blood supply to an organ is temporarily or permanently performed to minimize blood loss during a surgical procedure.

Additionally, there are disorders where the location of certain blood containing structures is important but not immediately obvious to surgeons during an operation. Knowledge of where those structures are is very important and could greatly improve the safety of various surgical procedures.

Patients of the investigator who are scheduled for foot surgery will be provided the opportunity to participate in this research. After giving informed consent, hyperspectral images will be obtained at various points during the surgical procedure.

As this technology is non-invasive, it is not expected to interfere with or change the procedure they are undergoing. Once the surgical procedure is complete, imaging will be saved to a disk for later evaluation.

100 subjects will participate in this study.

DETAILED DESCRIPTION:
The hyperspectral imager will be turned on at various time points during surgery, to measure the spectral wavelengths of tissues. The surgery being performed will in no way be altered by the imaging device and post surgical follow-up of patients will be standard of care appropriate to the surgical procedure.

Patients will have HSI performed only during their surgery. They will not receive additional medications and will have no additional follow up. Participating in this study will not add extra appointments, procedures, or time requirements for the patient. The patient's medical record may be referenced for information after the surgery for up to one year. There are no costs to the patient for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* 18 years or older undergoing foot surgery
* Speak and read English or Spanish.
* Able to provide written informed consent.

Exclusion Criteria:

* Patients unable to give written informed consent
* Patients who cannot speak and read English or Spanish will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the investigator scheduled for foot surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06-13 (Estimated); Primary Completion 2014-06-13 (Estimated); Study Completion 2015-06-13 (Actual)

PRIMARY OUTCOMES:
Correlation of HSI images with patient outcomes | 1 year
  Patient video images will be correlated with individual outcomes. Patients undergoing similar procedures will then be compared in terms of surgical outcome and differences in hyperspectral imaging variables.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Lavery, DPM, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas